CLINICAL TRIAL: NCT01116726
Title: Promoting Behavioral Change for Oral Health in American Indian Mothers and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-0894; 09-004E (Other Grant/Funding Number: National Institute of Dental and Craniofacial Research); 1U54DE019259 (NIH)
Record Dates: First submitted 2010-04-29; First posted 2010-05-05 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Early Childhood Dental Caries
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational interviewing and enhanced community services (Experimental): Motivational interviewing sessions will involve home visits concentrating on the mitigation of behavioral risk factors for early childhood caries, provided shortly after childbirth, and at 6, 12, and 18 months. Enhanced community services will involve development of culturally appropriate messages related to the mitigation of risk factors for ECC through public service announcements and brochures.
  Interventions: Behavioral: Motivational interviewing; Behavioral: Enhanced community services
- Enhanced community services (Active Comparator): Enhanced community services will involve development of culturally appropriate messages related to the mitigation of behavioral risk factors for early childhood caries through public service announcements and brochures.
  Interventions: Behavioral: Enhanced community services

INTERVENTIONS:
Behavioral: Motivational interviewing — MI sessions will involve home visits concentrating on the mitigation of behavioral risk factors for early childhood caries. These will take place shortly after childbirth and at months 6, 12, and 18.
  Arms: Motivational interviewing and enhanced community services
Behavioral: Enhanced community services — Enhanced community services will involve the development of culturally appropriate messages related to the mitigation of behavioral risk factors for early childhood caries through public service announcements and brochures.

SUMMARY:
A program of motivational interviewing plus enhanced community services in prevention of early childhood caries vs. enhanced community services alone for American Indian mothers and their children will reduce the childrens' decayed, missing, and filled tooth surfaces measure over a 3-year period.

DETAILED DESCRIPTION:
This is a randomized, controlled clinical trial. Six hundred mothers and their children will be randomized over a 2-year period to motivational interviewing (MI) plus enhanced community services vs. enhanced community services alone in equal numbers in the 2 groups. The MI sessions will involve home visits concentrating on the mitigation of behavioral risk factors for early childhood caries (ECC), shortly after childbirth and at 6, 12, and 18 months. The enhanced community services will involve development of culturally appropriate messages related to the mitigation of risk factors for ECC through public announcements and simple brochures. The primary outcome measure will be decayed, missing, and filled tooth surfaces (dmfs) of the children at ages 1, 2, and 3. Secondary outcomes will include children's ds, % with dmfs and ds >0, mother's dental knowledge, attitudes, and behaviors, caries patterns, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Be American Indian, as defined by the tribe
* Be mothers or caregivers of newborn children
* At least 15-44 years of age (Minors who are 15-17 years of age must get consent from a parent or legal guardian according to Tribal, State, and IHS rules and regulations)
* Able to read, understand, and sign a consent form/assent form,
* Be willing and able to follow study procedures and instructions.

Exclusion Criteria:

* No exclusion criteria. Although expected to be rare, if the father is a sole caregiver, he and his child will be eligible for the study.

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1134 (Actual)
Dates: Start 2011-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Decayed,missing, and filled tooth surfaces (dmfs) | Over 3 years

SECONDARY OUTCOMES:
Dental knowledge, attitudes, and behaviors of the mothers | Over 3 years
Dental caries patterns of the children | Over 3 years
Costs of dental care | Up to 3 years after randomization
Other decayed, missing, and filled tooth surfaces measures | Over 3 years
  ds, % of children with dmfs and ds >0

CONTACTS AND LOCATIONS:
Overall Officials: Terry Batliner, DDS, MBA, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Batliner T, Fehringer KA, Tiwari T, Henderson WG, Wilson A, Brega AG, Albino J. Motivational interviewing with American Indian mothers to prevent early childhood caries: study design and methodology of a randomized control trial. Trials. 2014 Apr 14;15:125. doi: 10.1186/1745-6215-15-125. PMID 24735707
- [Derived] Batliner TS, Tiwari T, Henderson WG, Wilson AR, Gregorich SE, Fehringer KA, Brega AG, Swyers E, Zacher T, Harper MM, Plunkett K, Santo W, Cheng NF, Shain S, Rasmussen M, Manson SM, Albino J. Randomized Trial of Motivational Interviewing to Prevent Early Childhood Caries in American Indian Children. JDR Clin Trans Res. 2018 Oct;3(4):366-375. doi: 10.1177/2380084418787785. Epub 2018 Jul 12. PMID 30238061
- [Derived] Albino J, Tiwari T, Gansky SA, Henshaw MM, Barker JC, Brega AG, Gregorich SE, Heaton B, Batliner TS, Borrelli B, Geltman P, Kressin NR, Weintraub JA, Finlayson TL, Garcia RI; Early Childhood Caries Collaborating Centers. The basic research factors questionnaire for studying early childhood caries. BMC Oral Health. 2017 May 19;17(1):83. doi: 10.1186/s12903-017-0374-5. PMID 28526003